CLINICAL TRIAL: NCT02118948
Title: Development of a Novel HIV Risk Reduction Intervention for Abused Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: University of Rochester (Other)
Responsible Party: Principal Investigator, Theresa E. Senn, Senior Research Scientist and Associate Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH095362 (NIH)
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Sexual Behavior
Keywords: abuse; sexual behavior; sexual risk reduction; behavioral intervention
MeSH Terms: conditions — Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Abuse-focused intervention (Experimental): Participants attend 5 weekly, 2-hour intervention sessions focused on the psychological consequences of abuse, current sexual risk behavior, and the link between the two.
  Interventions: Behavioral: Abuse-focused intervention
- Sexual behavior-focused intervention (Active Comparator): Participants attend 5 weekly, 2-hour intervention sessions focused on current sexual risk behavior.
  Interventions: Behavioral: Sexual behavior-focused intervention

INTERVENTIONS:
Behavioral: Abuse-focused intervention
  Arms: Abuse-focused intervention
Behavioral: Sexual behavior-focused intervention
  Arms: Sexual behavior-focused intervention

SUMMARY:
The purpose of this study is to develop and evaluate an HIV risk reduction intervention for women with a history of abuse.

DETAILED DESCRIPTION:
The purpose of the proposed research is to pilot test an innovative, theoretically-guided sexual risk reduction intervention for women with a history of abuse. T intervention builds on previous findings suggesting that it is important to address the psychological consequences of abuse, as well as the typical antecedents of sexual risk behavior. To inform intervention development, women who reported a history of abuse were recruited to participate in key informant interviews. Based on interview findings and guided by theory and empirical precedent, a novel sexual risk reduction intervention was developed and refined. The intervention will be pilot tested with 80 women recruited from a publicly-funded clinic who report a history of abuse and current sexual risk behavior. These women will complete a computerized survey to assess abuse, adult sexual risk behavior, HIV-related information, safer sex motivation, behavioral skills, interpersonal trust, guilt, and powerlessness. Behavioral skills will also be assessed through role-plays and simulation scenarios. Women will be randomly assigned to the novel intervention or to a structurally equivalent intervention focused only on the psychological antecedents of sexual risk behavior. Three months after intervention completion, women will return to complete computerized interviews and behavioral skills assessments. The long-term goal of this research is to develop a feasible and effective sexual risk reduction intervention for women who have a history of abuse.

ELIGIBILITY:
Inclusion Criteria:

* history of abuse
* current sexual risk behavior

Exclusion Criteria:

* less than age 18
* impaired mentally
* do not speak English
* severely depressed or suicidal
* HIV+

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
change in number of sexual partners in the past 3 months | baseline and 3 months
  at baseline and at 3 months post intervention, participants will respond to the question, "How many sexual partners have you had in the past 3 months?", assessed by computerized survey
change in number of episodes of unprotected sex in the past 3 months | baseline and 3 months
  at baseline and at 3 months post intervention, participants will report (a) the number of times they had sex with a primary partner in the past 3 months (b) out of the number of sex episodes with a primary partner in the past 3 months, how many times a condom was used; (c) the number of times they had sex with non-primary partners in the past 3 months; and (d) out of the number of sex episodes with a non-primary partner in the past 3 months, how many times a condom was used; responses to these 4 items will be used to determine the change in the total number of unprotected sex episodes (past 3 months) from baseline to 3 months post-intervention, assessed by computerized survey

SECONDARY OUTCOMES:
change in scores on the HIV Knowledge Questionnaire | baseline and 3 months
  assessed by computerized survey
change in scores on Condom Attitudes measure | baseline and 3 months
  condom attitudes measure assessing (a) attitudes towards condom use in primary relationships; (b) attitudes towards condom use in non-primary relationship; (c) pleasure-related condom attitudes; and (d) respect-related condom attitudes, assessed by computerized survey
change in performance on condom application exercise | baseline and 3 months
  participant is observed and scored while placing a condom on a model
change in scores on Traumatic Sexualization Survey | baseline and 3 months
  assessed by computerized survey
change in scores on Dyadic Trust Scale | baseline and 3 months
  assessed by computerized survey
change in scores on Abuse-Related Beliefs Questionnaire | baseline and 3 months
  assessed by computerized survey
change in scores on Sexual Relationship Power Scale | baseline and 3 months
  assessed by computerized survey
change in scoress on the PTSD Checklist-Civilian Version | baseline and after each intervention session
  assessed via computerized survey at baseline and via paper and pencil survey at the end of each intervention session

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States